CLINICAL TRIAL: NCT05493501
Title: A Randomized, Three-Arm, Open-Label Phase 3b Clinical Trial of Aumolertinib, Versus Aumolertinib With Chemotherapy, Versus Osimertinib for Patients With Metastatic NSCLC and an EGFR Mutation (TREBLE)
Brief Title: Aumolertinib With Chemotherapy or Alone Compared With Osimertinib in Patients With Epidermal Growth Factor Receptor-Mutant Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study is being closed based on corporate changes at EQRx and is not related to any efficacy or safety issues with aumolertinib.
Sponsor: EQRx International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EQ143-301; 2022-002674-93 (EudraCT Number)
Record Dates: First submitted 2022-06-24; First posted 2022-08-09 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2023-10

CONDITIONS: NSCLC
MeSH Terms: interventions — aumolertinib; osimertinib; Pemetrexed; Cisplatin; Carboplatin; Paclitaxel; Taxes; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Aumolertinib monotherapy (Experimental)
  Interventions: Drug: Aumolertinib monotherapy
- Aumolertinib + platinum-based doublet chemotherapy (Experimental): For adenocarcinoma, either:
  * Aumolertinib + cisplatin with pemetrexed, or
  * Aumolertinib + carboplatin with pemetrexed
  For squamous cell carcinoma, one of the following:
  * Aumolertinib + cisplatin or carboplatin with paclitaxel;
  * Aumolertinib + cisplatin or carboplatin with albumin-bound paclitaxel; or
  * Aumolertinib + cisplatin or carboplatin with gemcitabine
  Interventions: Drug: Aumolertinib monotherapy; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin; Drug: Paclitaxel; Drug: Nab paclitaxel; Drug: Gemcitabine
- Osimertinib monotherapy (Active Comparator)
  Interventions: Drug: Osimertinib monotherapy

INTERVENTIONS:
Drug: Aumolertinib monotherapy — Administered orally, once daily as two 55-mg tablets for a total dose of 110 mg.
  Other Names: EQ143, HS-10296
  Arms: Aumolertinib + platinum-based doublet chemotherapy; Aumolertinib monotherapy
Drug: Osimertinib monotherapy — 80 mg tablet administered orally, once daily
  Other Names: Tagrisso
  Arms: Osimertinib monotherapy
Drug: Pemetrexed — Administered by IV Infusion per prescribing information. Maybe be continued as maintenance therapy
  Other Names: Alimta
  Arms: Aumolertinib + platinum-based doublet chemotherapy
Drug: Cisplatin — Administered by IV Infusion given over 4 fixed cycles (q3wk × 4 cycles) per prescribing information.
  Arms: Aumolertinib + platinum-based doublet chemotherapy
Drug: Carboplatin — Administered by IV Infusion given over 4 fixed cycles (q3wk × 4 cycles) per prescribing information.
  Arms: Aumolertinib + platinum-based doublet chemotherapy
Drug: Paclitaxel — Administered by IV Infusion given over 4 -6 fixed cycles per prescribing information.
  Other Names: Taxol
  Arms: Aumolertinib + platinum-based doublet chemotherapy
Drug: Nab paclitaxel — Administered by IV Infusion given over 4 fixed cycles per prescribing information.
  Other Names: Abraxane; Albumin-bound paclitaxel
  Arms: Aumolertinib + platinum-based doublet chemotherapy
Drug: Gemcitabine — Administered by IV Infusion over 4 fixed cycles per prescribing information.
  Other Names: Gemzar
  Arms: Aumolertinib + platinum-based doublet chemotherapy

SUMMARY:
Aumolertinib is a third-generation epidermal growth factor receptor (EGFR) tyrosine kinase inhibitor (TKI) that targets EGFR mutations. The reason for this study is to learn whether adding chemotherapy to a new investigational drug called aumolertinib helps to slow or stop cancer growth in people with EGFR mutation-positive, locally advanced or metastatic non-small cell lung cancer (NSCLC). The study will compare this new combination of drugs to osimertinib, given alone. Aumolertinib given alone will also be used in the study, and it will be looked at in comparison with osimertinib given alone.

This is a randomized, open-label study with 3 different groups that are listed below. "Randomized" means the study treatment participants take will be chosen by chance (decided at random by a computer). "Open-label" means that the participant, the study doctor, and the Sponsor will know which study treatment each participant is receiving.

Participants will be randomly assigned to one of the following 3 treatment groups:

* Group 1: Treatment with aumolertinib alone, taken orally (by mouth) as a pill once a day. Around 100 participants will be randomly assigned to this group.
* Group 2: Treatment with aumolertinib taken orally as a pill once a day, in combination with chemotherapy given intravenously (IV; through a needle placed in a vein) on the schedule provided by the study doctor. Around 200 participants will be randomly assigned to this group.
* Group 3: Treatment with osimertinib alone, taken orally as a pill once a day. Around 200 participants will be randomly assigned to this group.

Because there will be twice as many participants in Group 2 and Group 3 as in Group 1, the chance of a participant being randomly assigned to either of those groups is twice as likely as being assigned to Group 1.

Participants can continue to receive study treatment as long as they have not withdrawn consent, as long as they choose to continue to receive study treatment and are judged by their doctor to continue to receive clinical benefit from receiving the study treatment, and as long as no other study treatment and/or study discontinuation criteria are met .

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 18 years of age (or the legal age of consent in the jurisdiction in which the study is taking place)
2. Has pathologically confirmed NSCLC that is Stage IIIB, metastatic (Stage IVA or IVB), or recurrent, and which is not amenable to curative intent therapy.
3. Tumor harbors one of the 2 common EGFR mutations known to be associated with EGFR-TKI sensitivity-ex19del or L858R-either alone or in combination with other EGFR mutations (eg, G719X, exon 20 insertions, S7681, L861Q)
4. Has Eastern Cooperative Oncology group performance status of 0, 1, or 2 at the time of enrollment.
5. Has adequate organ function at the time of enrollment.
6. Has QTc interval of ≤ 470 ms
7. Male participants must agree to use a highly effective method of contraception and to refrain from donating sperm while receiving study treatment
8. Female participants are eligible to participate if not pregnant or breastfeeding, and at least one of the following conditions applies: is not of childbearing potential OR is of childbearing potential and using a highly effective contraceptive method while receiving study treatment AND agrees not to donate eggs (ova, oocytes) during this period
9. All female participants must have a negative serum or urine pregnancy test result within 48 hours prior to initiation of study drug dosing

Exclusion Criteria:

1. Is a candidate for curative intent therapy for the NSCLC diagnosis.
2. Tumor has mixed small-cell and non-small-cell pathology.
3. Has received prior systemic treatment for metastatic NSCLC. Prior chemotherapy or immunotherapy is permitted, provided that it was used for treatment of locoregional NSCLC as a component of curative intent therapy and administration was completed more than 6 months ago.
4. Has refractory nausea and vomiting, chronic gastrointestinal disease(s), inability to swallow the formulated product (percutaneous endoscopic gastrostomy tube administration may be allowed if tablets are not crushed), or a history of previous significant bowel resection-any of which would preclude adequate absorption of aumolertinib or osimertinib.
5. Has active or past medical history of interstitial lung disease, drug-induced interstitial lung disease or radiation pneumonitis that required steroid treatment
6. Has evidence of active bacterial, viral, or fungal infection which would preclude safe enrollment, as assessed by the treating Investigator.
7. Has significant concomitant condition, that in the Investigator's judgment would prevent the participant from receiving study treatment or being followed in this study, or which otherwise renders the participant inappropriate for the study.
8. For participants in the aumolertinib monotherapy and aumolertinib with chemotherapy arms, use of strong CYP3A4 inhibitors/inducers within 14 days before initial study drug dosing and use of grapefruit-containing products within 72 hours before initial study drug dosing is prohibited.
9. Has a history of prolonged QT syndrome or Torsades de Pointes
10. Has any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG, including evidence of QT prolongation (QTc >470 ms for males and >480 ms for females) or has any factor, including any current medication(s), known to increase the risk of QTc prolongation or the risk of arrhythmic events
11. Hypersensitivity or allergy to aumolertinib or osimertinib or their excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Highlands Oncology Group, Springdale, Arkansas
  - Memorial Cancer Institute, Hollywood, Florida
  - Memorial Cancer Institute, Pembroke Pines, Florida
  - QCCA - Mission Blood & Cancer, Des Moines, Iowa
  - Summit Health, Florham Park, New Jersey
  - SCRI - Tennessee Oncology PLLC- Chattanooga, Chattanooga, Tennessee
  - SCRI - Tennessee Oncology- Nashville, Nashville, Tennessee
  - Northwest Medical Specialties, PLLC, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Aumolertinib + Platinum-based Doublet Chemotherapy: For adenocarcinoma, either:
  * Aumolertinib + cisplatin with pemetrexed, or
  * Aumolertinib + carboplatin with pemetrexed
  For squamous cell carcinoma, one of the following:
  * Aumolertinib + cisplatin or carboplatin with paclitaxel;
  * Aumolertinib + cisplatin or carboplatin with albumin-bound paclitaxel; or
  * Aumolertinib + cisplatin or carboplatin with gemcitabine
  Aumolertinib monotherapy: Administered orally, once daily as two 55-mg tablets for a total dose of 110 mg.
  Pemetrexed: Administered by IV Infusion per prescribing information. Maybe be continued as maintenance therapy
  Cisplatin: Administered by IV Infusion given over 4 fixed cycles (q3wk × 4 cycles) per prescribing information.
  Carboplatin: Administered by IV Infusion given over 4 fixed cycles (q3wk × 4 cycles) per prescribing information.
  Paclitaxel: Administered by IV Infusion given over 4 -6 fixed cycles per prescribing information.
  Nab paclitaxel: Administered by IV Infusion given over 4 fixed cycles per prescribing information.
  Gemcitabine: Administered by IV Infusion over 4 fixed cycles per prescribing information.
Period: Overall Study
Arm/Group | Aumolertinib Monotherapy | Aumolertinib + Platinum-based Doublet Chemotherapy | Osimertinib Monotherapy
Started | 1 | 2 | 5
Completed | 0 | 0 | 0
Not Completed | 1 | 2 | 5

BASELINE CHARACTERISTICS:
Population: Study terminated early, no participants completed the study, no participants were analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aumolertinib Monotherapy | Aumolertinib + Platinum-based Doublet Chemotherapy | Osimertinib Monotherapy | Total
Number analyzed (Participants) | 1 | 2 | 5 | 8
Age, Continuous [Mean (Full Range); unit: years] | 69 [69 to 69] | 71 [66 to 75] | 63 [52 to 74] | 66 [52 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 4 | 7
  Male | 0 | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 1 | 2 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 1 | 2 | 5 | 8
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) as Assessed by Blinded Independent Central Review (BICR) Per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: PFS is defined as the time from date of randomization until date of disease progression or death due to any cause, whichever occurs first.
Time Frame: Up to 5 years
Population: data not collected, 0 participants analyzed
Arm/Group | Aumolertinib Monotherapy | Aumolertinib + Platinum-based Doublet Chemotherapy | Osimertinib Monotherapy
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from date of randomization until death from any cause.
Time Frame: Up to 6 years
Population: data not collected, 0 participants analyzed
Arm/Group | Aumolertinib Monotherapy | Aumolertinib + Platinum-based Doublet Chemotherapy | Osimertinib Monotherapy
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Objective Response Rate (ORR) as Assessed by BICR Per RECIST v1.1
Description: ORR is defined as proportion of participants who achieve a complete response or partial response at any time before progressive disease or initiating a subsequent anticancer therapy.
Time Frame: Up to 5 years
Population: data not collected, 0 participants analyzed
Arm/Group | Aumolertinib Monotherapy | Aumolertinib + Platinum-based Doublet Chemotherapy | Osimertinib Monotherapy
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Disease Control Rate (DCR) as Assessed by BICR Per RECIST v1.1
Description: DCR is defined as the proportion of participants who have a best overall response of complete response or partial response or stable disease.
Time Frame: Up to 5 years
Population: data not collected, 0 participants analyzed
Arm/Group | Aumolertinib Monotherapy | Aumolertinib + Platinum-based Doublet Chemotherapy | Osimertinib Monotherapy
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Tumor Growth Rate (TGR) as Assessed by BICR Per RECIST v1.1
Description: TGR is defined as the constant exponential growth rate estimated using the sum of longest diameters based on radiological tumor assessment per RECIST v1.1.
Time Frame: Up to 5 years
Population: data not collected, 0 participants analyzed
Arm/Group | Aumolertinib Monotherapy | Aumolertinib + Platinum-based Doublet Chemotherapy | Osimertinib Monotherapy
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Duration of Response (DOR) as Assessed by BICR Per RECIST v1.1
Description: DOR is defined as date of first response (complete response or partial response) until date of disease progression or death due to any cause, whichever occurs first
Time Frame: Up to 5 years
Population: data not collected, 0 participants analyzed
Arm/Group | Aumolertinib Monotherapy | Aumolertinib + Platinum-based Doublet Chemotherapy | Osimertinib Monotherapy
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Depth of Response (DepOR) as Assessed by BICR Per RECIST v1.1
Description: DepOR is defined as the relative change in target lesion tumor size (calculated as the sum of the longest diameters of the target lesions, in the absence of new lesions or progression of nontarget lesions) as compared to baseline.
Time Frame: Up to 5 years
Population: data not collected, 0 participants analyzed
Arm/Group | Aumolertinib Monotherapy | Aumolertinib + Platinum-based Doublet Chemotherapy | Osimertinib Monotherapy
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: PFS as Assessed by the Investigator Per RECIST v1.1
Description: as for outcome 1
Time Frame: Up to 5 years
Population: data not collected, 0 participants analyzed
Arm/Group | Aumolertinib Monotherapy | Aumolertinib + Platinum-based Doublet Chemotherapy | Osimertinib Monotherapy
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: ORR as Assessed by the Investigator Per RECIST v1.1
Description: ORR is defined as the proportion of participants who achieve a complete response or partial response at any time before disease progression or initiating a subsequent anticancer therapy.
Time Frame: Up to 5 years
Population: data not collected, 0 participants analyzed
Arm/Group | Aumolertinib Monotherapy | Aumolertinib + Platinum-based Doublet Chemotherapy | Osimertinib Monotherapy
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: DCR as Assessed by the Investigator Per RECIST v1.1
Description: as for outcome 4
Time Frame: Up to 5 years
Population: data not collected, 0 participants analyzed
Arm/Group | Aumolertinib Monotherapy | Aumolertinib + Platinum-based Doublet Chemotherapy | Osimertinib Monotherapy
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: TGR as Assessed by the Investigator Per RECIST v1.1
Description: as for outcome 5
Time Frame: Up to 5 years
Population: data not collected, 0 participants analyzed
Arm/Group | Aumolertinib Monotherapy | Aumolertinib + Platinum-based Doublet Chemotherapy | Osimertinib Monotherapy
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: DOR as Assessed by the Investigator Per RECIST v1.1
Description: DOR is defined as date of first response (complete response or partial response) until the date of disease progression or death due to any cause, whichever occurs first.
Time Frame: Up to 5 years
Population: data not collected, 0 participants analyzed
Arm/Group | Aumolertinib Monotherapy | Aumolertinib + Platinum-based Doublet Chemotherapy | Osimertinib Monotherapy
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: DepOR as Assessed by the Investigator Per RECIST v1.1
Description: as for outcome 7
Time Frame: Up to 5 years
Population: data not collected, 0 participants analyzed
Arm/Group | Aumolertinib Monotherapy | Aumolertinib + Platinum-based Doublet Chemotherapy | Osimertinib Monotherapy
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Quality of Life as Assessed by the National Cancer Institute Patient Reported Outcomes Common Terminology Criteria for Adverse Events (NCI PRO-CTCAE) Questionnaire
Description: NCI PRO-CTCAE questionnaire responses are scored from 0 to 4, wherein lower values represent a better outcome. For this trial, the burden of symptoms that will be captured by this questionnaire comprises nausea, diarrhea, and rash.
Time Frame: Up to 5 years
Population: data not collected, 0 participants analyzed
Arm/Group | Aumolertinib Monotherapy | Aumolertinib + Platinum-based Doublet Chemotherapy | Osimertinib Monotherapy
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Rate of Circulating Tumor DNA (ctDNA) Clearance
Description: ctDNA clearance is defined as when a detectable EGFR mutation in ctDNA at baseline becomes undetectable or drops below a predetermined threshold. Rate of ctDNA clearance is defined as 100 × number of participants who are ctDNA-negative at 6 weeks divided by number of participants who are ctDNA-positive at baseline.
Time Frame: 6 weeks
Population: data not collected, 0 participants analyzed
Arm/Group | Aumolertinib Monotherapy | Aumolertinib + Platinum-based Doublet Chemotherapy | Osimertinib Monotherapy
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Plasma Concentration of Aumolertinib
Description: Plasma concentration is defined as the measured drug concentration of aumolertinib.
Time Frame: Up to approximately 5 months
Population: data not collected, 0 participants analyzed
Arm/Group | Aumolertinib Monotherapy | Aumolertinib + Platinum-based Doublet Chemotherapy | Osimertinib Monotherapy
Number analyzed (Participants) | 0 | 0 | 0

17. Secondary Outcome: Plasma Concentration of Aumolertinib Metabolite
Description: Plasma concentration is defined as the measured drug concentration of aumolertinib metabolite.
Time Frame: Up to approximately 5 months
Population: data not collected, 0 participants analyzed
Arm/Group | Aumolertinib Monotherapy | Aumolertinib + Platinum-based Doublet Chemotherapy | Osimertinib Monotherapy
Number analyzed (Participants) | 0 | 0 | 0

18. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: This outcome will evaluate the incidence of participants with TEAEs, graded according to NCI CTCAE V5.
Time Frame: From date of treatment initiation until discontinuation from treatment (plus 28 days for TEAEs), up to 5 years
Population: data not collected, 0 participants analyzed
Arm/Group | Aumolertinib Monotherapy | Aumolertinib + Platinum-based Doublet Chemotherapy | Osimertinib Monotherapy
Number analyzed (Participants) | 0 | 0 | 0

19. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: This outcome will evaluate incidence of participants with SAEs, be graded according to NCI CTCAE V5.
Time Frame: From date of treatment initiation until discontinuation from treatment (plus 28 days for TEAEs), up to 5 years
Population: data not collected, 0 participants analyzed
Arm/Group | Aumolertinib Monotherapy | Aumolertinib + Platinum-based Doublet Chemotherapy | Osimertinib Monotherapy
Number analyzed (Participants) | 0 | 0 | 0

20. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: This outcome will evaluate incidence of participants with ECG abnormalities
Time Frame: From date of treatment initiation until discontinuation from treatment (plus 28 days for TEAEs), up to 5 years
Population: data not collected, 0 participants analyzed
Arm/Group | Aumolertinib Monotherapy | Aumolertinib + Platinum-based Doublet Chemotherapy | Osimertinib Monotherapy
Number analyzed (Participants) | 0 | 0 | 0

21. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: This outcome will evaluate incidence of participants with laboratory abnormalities, graded according to NCI CTCAE V5.
Time Frame: From date of treatment initiation until discontinuation from treatment (plus 28 days for TEAEs), up to 5 years
Population: data not collected, 0 participants analyzed
Arm/Group | Aumolertinib Monotherapy | Aumolertinib + Platinum-based Doublet Chemotherapy | Osimertinib Monotherapy
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected until the study reached early termination. Adverse events were collected from date of treatment initiation until discontinuation from treatment (plus 28 days for TEAEs), approximately 8 months, 17 days.
Description: The trial was discontinued at 8 months. No patients were analyzed.
Arm/Group | Aumolertinib Monotherapy | Aumolertinib + Platinum-based Doublet Chemotherapy | Osimertinib Monotherapy
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2 | 0/5
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2 | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aumolertinib Monotherapy (N=1) | Aumolertinib + Platinum-based Doublet Chemotherapy (N=2) | Osimertinib Monotherapy (N=5)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 3
Gastro-oesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 2 | 1
Skin Infection (Infections and infestations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 2
Hypotension (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-05-19): https://cdn.clinicaltrials.gov/large-docs/01/NCT05493501/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-16): https://cdn.clinicaltrials.gov/large-docs/01/NCT05493501/SAP_001.pdf